CLINICAL TRIAL: NCT04760171
Title: An ex Vivo Study to Purify Amyloid Fibrils and Solve Their 3D Structures Using Amyloid Proteins From Medullary Thyroid Cancer and Laryngeal Amyloidosis
Brief Title: Amyloid Proteins From Medullary Thyroid Cancer and Laryngeal Amyloidosis
Status: Not yet recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: EN21/138414
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Amyloid; Medullary Thyroid Cancer; Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Carcinoma, Medullary; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Excess tumour tissue resected from patients with known medullary thyroid cancer, or, laryngeal amyloidosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients diagnosed with medullary thyroid cancer (MTC) who are undergoing standard surgical treatment for their disease. This will be either hemithyroidectomy or total thyroidectomy. Patients with laryngeal amyloidosis (LA) who are undergoing standard surgical treatment of this disease. This will be microlaryngoscopy & biopsy/debulking

SUMMARY:
Using excess tumour samples that contain amyoid, from patients with Medullary Thyroid Cancer, we aim to determine the structures of ex vivo amyloid fibrils from human tumour tissue samples and compare them with that of existing stock of in vitro formed amyloid fibrils. This will permit the analysis of the effects of gene mutation and post-translational modification on the development of amyloid from a disease state.

Amyloid is known to accumulate in the brain tissue of patients with neuro-degenerative conditions such as Alzheimer's disease and Dementia. Therefore solving the structure of amyloid fibrils may aid the development of future treatments for these conditions.

DETAILED DESCRIPTION:
This is an anonymous, voluntary inclusion, laboratory based, basic science research study. Appropriate patients who meet the inclusion criteria and complete the consent process will be asked to donate a small sample of excess tumour tissue after the completion of their surgical procedure. This tissue will be transferred to the research laboratory in Leeds University for analysis and subject to a variety of investigations and scientific procedures to achieve the study objectives.

These include:

1. - amyloid extraction by tissue homogenization and centrifugation as already documented in the literature.
2. - mass spectrometry analysis to identify and characterize the most prominent proteins present in the amyloid deposits and their possible post-translational modifications.
3. - Transmission Electron Microscopy to characterize at the gross features of the extracted amyloid fibrils at low resolution (>20Å). This relatively simple procedure allows for quick characterization of the samples in order to optimize them for Atomic Force Microscopy (AFM) and Cryo-Electron Microscopy (Cryo-EM).
4. - Atomic Force microscopy to characterize helical parameters of the amyloid fibrils needed to calculate the structure from Cryo-EM data.
5. - Cryo-Electron Microscopy to elucidate the structure of the amyloids extracted from tissue affected in each disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with known or suspected MTC or LA
* Age >= 18 years, no upper age limit
* Able to provide informed consent for both surgical treatment and inclusion into this study
* For MTC patients, treatment recommendation from the Thyroid MDT is for either hemithyroidectomy or total thyroidectomy
* for LA patients, agreement with their attending clinician to undergo surgical debulking of disease under general anaesthetic. The procedure is called 'microlaryngoscopy and biopsy/debulking'

Exclusion Criteria:

* No known or suspected diagnosis of MTC or LA
* Age <18 years

  * Unable to provide informed consent
  * Treatment recommendation from Thyroid MDT is for any treatment excluding primary surgery (ie palliation, best supportive care, chemotherapy, radiotherapy etc)
  * For LA patients, no agreement between patient and attending clinician to proceed with surgery as primary treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with MTC, who have been recommended via the Thyroid Multi-Disciplinary team meeting, to undergo hemi or total thyroidectomy surgery.
  Patients with LA, who agree with their surgeon, to undergo surgical treatment of that condition
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Amyloid extraction by tissue homogenization and centrifugation | 12-24 months
  A standard laboratory technique for subsequent analysis
Transmission electron microscopy | 12-24 months
  To characterize the gross features of the extracted amyloid fibrils at low resolution (>20Å). This relatively simple procedure allows for quick characterization of the samples in order to optimize them for Atomic Force Microscopy (AFM) and Cryo-Electron Microscopy (Cryo-EM).
Atomic force microscopy | 12-24 months
  To characterize helical parameters of the amyloid fibrils needed to calculate the structure from Cryo-EM data.
Cryo-electron microscopy (Cryo-EM) | 12-24 months
  To elucidate the structure of the amyloids extracted from tissue affected in each disease
Mass spectrometry | 12-24 months
  Analysis to identify and characterize the most prominent proteins present in the amyloid deposits and their possible post-translational modifications.

CONTACTS AND LOCATIONS:
Overall Officials: James Moor, FRCS, Principal Investigator — Leeds Teaching Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
Samples will be anonymised, and research outputs will be based on the whole cohort. Therefore IPD will not be available.

REFERENCES:
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Knowles TP, Vendruscolo M, Dobson CM. The amyloid state and its association with protein misfolding diseases. Nat Rev Mol Cell Biol. 2014 Jun;15(6):384-96. doi: 10.1038/nrm3810. PMID 24854788
- [Background] Gallardo R, Iadanza MG, Xu Y, Heath GR, Foster R, Radford SE, Ranson NA. Fibril structures of diabetes-related amylin variants reveal a basis for surface-templated assembly. Nat Struct Mol Biol. 2020 Nov;27(11):1048-1056. doi: 10.1038/s41594-020-0496-3. Epub 2020 Sep 14. PMID 32929282
- [Background] Gallardo R, Ranson NA, Radford SE. Amyloid structures: much more than just a cross-beta fold. Curr Opin Struct Biol. 2020 Feb;60:7-16. doi: 10.1016/j.sbi.2019.09.001. Epub 2019 Nov 1. PMID 31683043